CLINICAL TRIAL: NCT00198549
Title: Phase IV Post-Approval Evaluation of Vitrase as an Adjuvant to Increase the Absorption and Dispersion of Other Injected Anesthetics for Ophthalmic Surgical Procedures
Brief Title: Evaluation of Vitrase as an Adjuvant to Increase Absorption and Dispersion of Other Injected Anesthetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISTA-VIT-SA-MA02
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Pain
Keywords: Adjuvants, Anesthesia; hyaluronate lyase
MeSH Terms: conditions — Pain | interventions — Chondroitinases and Chondroitin Lyases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vitrase (ovine hyaluronidase) Lyophilized

SUMMARY:
The purpose of this study is to evaluate Vitrase as an adjuvant to increase absorption and dispersion of other injected anesthetics

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an ophthalmic surgical procedure

Exclusion Criteria:

* Known allergy to bee venom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-09; Primary Completion 2005-01 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
To evaluate physician acceptance of efficacy of Vitrase as an adjuvant to increase absorption and dispersion of anesthetics used for ophthalmic surgical procedures

SECONDARY OUTCOMES:
To determine physician usage of and satisfaction with Vitrase in the 6200 USP unit vial

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Grillone, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- Cincinnati Eye Institute, Cincinnati, Ohio, United States